CLINICAL TRIAL: NCT00003420
Title: A Study of CT Scan Frequency in Patients With Stage I Testicular Teratoma
Brief Title: CT Scans in Treating Patients With Stage I Testicular Cancer After Undergoing Orchiectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Diagnostic
Other Study IDs: CDR0000066440; MRC-TE08; EU-98007; ISRCTN56475197
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2002-12

CONDITIONS: Testicular Germ Cell Tumor
Keywords: stage I malignant testicular germ cell tumor; testicular teratoma
MeSH Terms: conditions — Testicular Germ Cell Tumor; Testicular Neoplasms; Teratoma, Testicular

INTERVENTIONS:
Procedure: computed tomography

SUMMARY:
RATIONALE: Imaging procedures such as CT scans help the doctor in detecting cancer or the recurrence of cancer. Increasing the number of times a CT scan is given may improve the ability to detect stage I testicular cancer.

PURPOSE: Randomized clinical trial to determine if there is a different result from two different schedules of CT scans in treating patients with stage I testicular cancer after undergoing orchiectomy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether there is a difference between two schedules of CT scan surveillance in respect to stage of disease at relapse, survival, the investigation determining relapse, and incidence of second malignancies in patients with stage I testicular teratoma after orchidectomy.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center and presence of vascular invasion.

After orchidectomy, patients are randomized into two schedules (arms I and II) of CT scan follow up.

* Arm I: Patients repeat chest and abdominal CT scans no later than 3 months after orchidectomy and again at 12 months to confirm that the patient is clear of disease.
* Arm II: Patients repeat chest and abdominal CT scans at 3, 6, 9, 12, and 24 months after orchidectomy.

Patients are followed monthly for the first year after orchidectomy, then every 2 months for the second year, then every 3 months for the third year, and then every 4-6 months thereafter.

PROJECTED ACCRUAL: There will be 400-900 patients accrued into this study over 3-6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed nonseminomatous germ cell tumor of the testis Stage I disease:

  * No evidence of metastatic disease on clinical examination
  * Normal chest x-ray
  * Normal chest and abdominal CT scan
  * Normal serum tumor marker (AFP, HCG) after orchidectomy
* High risk patients should be considered for ongoing studies of adjuvant chemotherapy after orchidectomy, but those choosing not to take this option may enter this study
* Orchidectomy no greater than 8 weeks prior to randomization into this study

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other concurrent or prior malignancy except successfully treated nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 1997-07; Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon J.S. Rustin, MD, Study Chair — Mount Vernon Cancer Centre at Mount Vernon Hospital
Locations (1):
- Mount Vernon Hospital, Northwood, England, United Kingdom

REFERENCES:
- [Result] Rustin GJ, Mead GM, Stenning SP, Vasey PA, Aass N, Huddart RA, Sokal MP, Joffe JK, Harland SJ, Kirk SJ; National Cancer Research Institute Testis Cancer Clinical Studies Group. Randomized trial of two or five computed tomography scans in the surveillance of patients with stage I nonseminomatous germ cell tumors of the testis: Medical Research Council Trial TE08, ISRCTN56475197--the National Cancer Research Institute Testis Cancer Clinical Studies Group. J Clin Oncol. 2007 Apr 10;25(11):1310-5. doi: 10.1200/JCO.2006.08.4889. PMID 17416851
- [Result] Mead GM, Rustin GJ, Stenning SP, et al.: Medical Research Council trial of 2 versus 5 CT scans in the surveillance of patients with stage I non-seminomatous germ cell tumours of the testis. [Abstract] J Clin Oncol 24 (Suppl 18): A-4519, 221s, 2006.